CLINICAL TRIAL: NCT07366216
Title: The Effect of Different Dual-Task Conditions on Chewing Function in Individuals With Multiple Sclerosis
Brief Title: Chewing Under Dual-Tasking in MS
Status: Not yet recruiting | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Seda Nur Kemer, Principal investigator, PT, PhD, Ondokuz Mayıs University
Other Study IDs: 1919B012411772
Record Dates: First submitted 2026-01-09; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple Sclerosis
- Healthy Control

SUMMARY:
This study aims to investigate the effects of visual, auditory, and motor dual-task conditions on chewing performance in individuals with multiple sclerosis, compared with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 65 years
* Mini-Mental State Examination (MMSE) score of 24 or higher
* Right-hand dominance

Exclusion Criteria:

* Presence of visual and/or hearing impairment
* Presence of difficulties in solid food intake and/or complaints related to mastication
* Presence of neurological, psychological, cognitive, and/or chronic conditions that may affect mastication or chewing function
* History of interventions affecting oral structure (e.g., oral/maxillofacial surgery or radiotherapy) within the last month
* Known allergy to the food used in the test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consisted of individuals with multiple sclerosis and age-matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Test of Masticating and Swallowing Solids | Baseline (single-task and dual-task conditions assessed on the same day)
  Test of Masticating and Swallowing Solids (TOMASS) is a standardized clinical assessment used to evaluate solid bolus mastication and swallowing performance.
Mini-Mental State Examination (MMSE) | Baseline
  The MMSE is a brief, widely used screening tool for assessing global cognitive function.
Go/No-Go Test | Baseline (single-task and dual-task conditions assessed on the same day)
  The Go/No-Go Test is a neuropsychological assessment used to evaluate response inhibition and sustained attention.
Auditory Reaction Time Test | Baseline (single-task and dual-task conditions assessed on the same day)
  The Auditory Reaction Time Test is used to assess auditory attention and the speed of motor response to auditory stimuli.
Tap Tool | Baseline (single-task and dual-task conditions assessed on the same day)
  The Tap Tool is a neuropsychological and motor performance assessment used to evaluate psychomotor speed and fine motor control.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayis University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No